CLINICAL TRIAL: NCT00283517
Title: Electronic Schizophrenia Treatment Adherence Registry, eSTAR
Brief Title: A Registry of Treatment Adherence for Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Country Medical Director, Janssen-Cilag S.A., Spain
Other Study IDs: CR005548
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: Risperidone long-acting injection; Antipsychotic medication; Schizophrenia; Treatment retention; Observational study
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Antipsychotic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Drug: antipsychotics

INTERVENTIONS:
Drug: antipsychotics — as prescribed

SUMMARY:
The purpose of the study is to assess demographic, treatment, and outcome data in schizophrenia patients receiving treatment with long-acting injectable, tablet, or liquid formulations of first generation (conventional) or second generation (atypical) antipsychotic medications.

DETAILED DESCRIPTION:
Recent studies have suggested the superior effectiveness of second generation (atypical) antipsychotic medications over first generation (conventional) antipsychotics in preventing relapse during the treatment of schizophrenia. It is estimated that a majority of patients with schizophrenia have difficulty adhering to the daily regimen of oral medications, and the use of long-acting injectable antipsychotics has been shown to increase compliance. This study includes both retrospective and prospective observations of the treatments and outcomes associated with antipsychotic drug therapy as well as characteristics of the patient population. The study is not product specific and includes patients using therapy with long-acting injectable, tablet, or liquid formulations of conventional or atypical antipsychotic medications. All patients who enroll in the study start treatment with a new antipsychotic medication, which is to be used according to the product labeling in the local country. Retrospective data, collected over a minimum of 12 months, include patient diagnosis, age, sex, history of treatment with antipsychotic medications, hospitalization, Clinical Global Impression of severity of disease (CGI-severity), Global Assessment of Functioning (GAF), and the reason for starting a new antipsychotic treatment. Prospective data, collected every 3 months over 2 years, are evaluated to assess the effectiveness of treatment and include the patient's adherence to antipsychotic medication, CGI-severity, GAF, and clinical deterioration of the patient's condition. The study investigator enters the data into a registry either electronically or on paper record forms. Safety assessments include the incidence, type and severity of adverse events throughout the prospective phase of the study. Atypical or conventional antipsychotics, as tablet, liquid or injectable formulations as prescribed

ELIGIBILITY:
Inclusion Criteria:

* Patients starting treatment with a new antipsychotic medication, in accordance with product labeling in the local country
* Permitted by their physician and by the patient to participate in a clinical trial

Exclusion Criteria:

* Patients not meeting all of the inclusion criteria for entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients starting treatment with a new antipsychotic medication, in accordance with product labeling in the local area; permitted by their physician to participate in a clinical trial
Sampling Method: Non-Probability Sample
Enrollment: 2046 (Actual)
Dates: Start 2003-09; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To assess demographic, treatment, and outcome data in schizophrenia patients receiving treatment with long-acting injectable, tablet, or liquid formulations of first generation (conventional) or second generation (atypical) antipsychotics medications. | every 3 months over 2 years

SECONDARY OUTCOMES:
Safety assessments include the incidence, type and severity of adverse events throughout the prospective phase of the study. | every 3 months over 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.

REFERENCES:
- [Derived] Lambert T, Emmerson B, Hustig H, Resseler S, Jacobs A, Butcher B; e-STAR Research Group. Long acting risperidone in Australian patients with chronic schizophrenia: 24-month data from the e-STAR database. BMC Psychiatry. 2012 Mar 26;12:25. doi: 10.1186/1471-244X-12-25. PMID 22448928